CLINICAL TRIAL: NCT00372177
Title: The Use of Anti-CD4 mAb-Fragment for the Imaging of Chronic Inflammation in Patients With Active Rheumatoid Arthritis (an Open Proof of Concept Study)
Brief Title: The Use of Anti-CD4 Monoclonal Antibody (mAb)-Fragment for the Imaging of Chronic Inflammation in Patients With Active Rheumatoid Arthritis
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Biotectid GmbH (Industry)
Collaborators: Technische Universität Dresden (Other); University of Leipzig (Other)
Responsible Party: Biotectid GmbH, Biotectid GmbH
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: Biotectid POC EP 1645; EP 1645
Record Dates: First submitted 2006-09-05; First posted 2006-09-06 (Estimated); Last update posted 2008-05-28 (Estimated); Status verified 2008-05

CONDITIONS: Rheumatoid Arthritis; Polyarthritis; Rheumatism; Autoimmune Disease; Inflammation
Keywords: monoclonal antibody; diagnostics; RA; Immunoglobulins; molecular target; Tc99m-pertechnetate; Fab-fragment of Anti-human CD4; Radiopharmaceutical; chronic inflammatory diseases; active Rheumatoid Arthritis
MeSH Terms: conditions — Arthritis, Rheumatoid; Arthritis; Rheumatic Diseases; Autoimmune Diseases; Inflammation

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- EP1645 (Active Comparator): Single-Dose
  Interventions: Radiation: Fab-fragment of Anti-human CD4

INTERVENTIONS:
Radiation: Fab-fragment of Anti-human CD4 — Sterile lyophilized Powder for Preparation of a Solution and sterile labelling Buffer labelling with Tc99m-Pertechnetat Intravenous injection

SUMMARY:
Rheumatoid arthritis (RA) is a disease with a large economic impact due to the long lasting disabling nature of the disease. Furthermore, diagnosis of the disease is difficult and only a scheme with different symptoms is used to diagnose rheumatoid arthritis, often only by probability.

Due to the fact that effective disease modifying pharmacological treatment is available and should be started early in established cases of RA, in combination with the adverse effect potential of these substances (e.g. methotrexate), a fast reliable diagnostic tool to diagnose rheumatoid arthritis would be highly appreciated by the medical community and the patients. Furthermore, for invasive treatments (surgery, puncture), an imaging method to display the activity pattern in different joints would be a major advantage.

For the evaluation of the effectiveness of pharmacological therapy in rheumatoid arthritis, up to now, radiological measurements of the destruction process of the joints are used. This method has the disadvantage that it is time consuming insofar as changes in the radiological images must occur. It allows only an evaluation if the joints are destructed (which should be excluded by the new therapy regimen). Again, a quantifiable method for the determination of the effects of new therapeutic approaches would be highly appreciated.

DETAILED DESCRIPTION:
The substance will be used as iv injection due to the protein nature of the antibody and, to ensure a fast distribution within the body. The study will be performed as an open clinical trial due to the fact that the applied radiation has to be documented; the use of "placebo" radiation would be unethical.

It is expected, that the new antibody fragment with its radioactive linkage will display an image of the activity distribution of the disease. Due to the fact that only patients with active disease have to be imaged and, to allow for comparison of the activity and the clinical distribution of the disease, this proof of concept study (phase I study) will be performed in patients with active disease. Healthy volunteers could not display an activity pattern of the disease. Furthermore, it seems to be unethical to use volunteers for studies with radioactivity with such a risk/benefit ratio (radiation risks vs. missing chance of display of tissue distribution) in a proof of concept study.

ELIGIBILITY:
Inclusion Criteria:

* Male and female subjects above 50 years of age
* Suffering from joint pain which is due to active rheumatoid arthritis
* Obvious signs of inflammation in at least one joint (e.g. swelling, erythema, or local elevated temperature)
* Otherwise healthy
* Informed consent

Exclusion Criteria:

* Patients 80 years and older
* Clinically significant disease of the cardiovascular system, respiratory system, hepato-biliary system or central nervous system (CNS)
* Excretory hepatic or renal insufficiency
* Regular intake of any drug, except for hormone replacement therapy in females
* Previous administration of xenogenous proteins
* History of anaphylactic reaction to any drug administered by a parenteral pathway
* Previous participation in a radiopharmaceutical drug trial (unless the effective dose acquired by participation in the current trial will remain below 10 mSv)
* Participation in any clinical drug trial within 3 months prior to enrolment
* Women of child-bearing potential (child-bearing potential to be ruled out by one of the following: at least 2 years past menopause, hysterectomy, bilateral oophorectomy, or bilateral tubal ligation)
* Long term medication with strong antiphlogistic agents/pain killers such as methotrexate, corticoids, or immunosuppressants prior to enrolment

Ages: 50 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 5 (Actual)
Dates: Start 2007-07; Primary Completion 2008-05 (Actual); Study Completion 2008-05 (Actual)

PRIMARY OUTCOMES:
safety and tolerability of this diagnostic agent | duration of study

SECONDARY OUTCOMES:
endpoint for the proof of concept will be the number of patients needed to obtain a series of equal results | duration of study

CONTACTS AND LOCATIONS:
Overall Officials: Osama Sabri, Prof. Dr., Principal Investigator — Clinic and Policlinic for Nuclear Medicine, Medical Faculty, University of Leipzig, Germany
Locations (1):
- Clinic and Policlinic for Nuclear Medicine, Medical faculty, University of Leipzig, Leipzig, Saxony, Germany

REFERENCES:
- See also: Related Info — http://nuklmed.uniklinikum-leipzig.de/